CLINICAL TRIAL: NCT02440282
Title: Comparison of Anesthetic Modalities on Hemodynamic Stability and Postoperative Pain in Diabetic Foot Patients Undergoing Minor Lower Extremity Amputation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-1022
Record Dates: First submitted 2015-04-24; First posted 2015-05-12 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Diabetic Foot Ulcer; Lower Extremity Amputation
Keywords: patients
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: patients undergo general anesthesia
- Group B: spinal anesthesia
- Group C: ultrasound-guided sciatic nerve block

SUMMARY:
Diabetic foot ulcer is the most common cause of non traumatic lower extremity amputations (LEA) associated with diabetes. Traditionally general and spinal anesthesia were the preferred modality of anesthesia. The use of sciatic nerve block has recently gained popularity, however, without the supporting evidence of any benefits. This study was to evaluate the comparison of anesthesia modalities for hemodynamic stability and postoperative pain in diabetic foot patients undergoing minor LEA.

ELIGIBILITY:
Inclusion Criteria:

* diabetic foot patients who underwent minor LEA

Exclusion Criteria:

* emergency cases
* patients who underwent major upper or lower extremity amputations
* patients who received general anesthesia following fail regional or spinal anesthesia
* patients who underwent LEA within 1year, and patients who underwent other concomitant surgeries

Ages: 29 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive 86 diabetic foot patients who underwent minor LEA
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure | every ten minutes from preinduction to 30minutes after sugery
Mean blood pressure | from arrival at recovery room until 20miutes after surgery at recovery room
Heart rate | every ten minutes from preinduction to 30minutes after sugery
Heart rate | from arrival at recovery room until 20miutes after surgery at recovery room